CLINICAL TRIAL: NCT06207669
Title: The Effect of Music Therapy on Itching, Muscle Cramps and Comfort in Individuals Receiving Hemodialysis Treatment
Brief Title: Music Therapy for Individuals Receiving Hemodialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Soner Telli, master student, Amasya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: amasyau-soner_1
Record Dates: First submitted 2023-12-27; First posted 2024-01-17 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy group (Experimental): A musical concert will be held for the participants in the Hicaz makam.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — Music therapy will be applied to individuals in the clinic for 30 minutes after the 2nd hour of each hemodialysis session for 4 weeks.

SUMMARY:
There are studies in the world where music therapy is used in the management of symptoms in hemodialysis, but the number of studies in our country is insufficient. This study will be carried out to determine the effect of music therapy on itching, muscle cramps and comfort level in individuals receiving hemodialysis HD treatment.

The research will be conducted in the Amasya Sabuncuoğlu Şerefeddin Training and Research Hospital Dialysis Unit Hemodialysis Clinic, with a pre-test post-test single group, quasi-experimental research design. The sample of the research; It will constitute 38 individuals aged 18 and over who have been receiving hemodialysis treatment for at least 6 months. Music therapy will be applied to the participants in the clinic for 30 minutes after the 2nd hour of each hemodialysis session for 4 weeks.

Research data will be collected between January and March 2024 using the Introductory Information Form, 5-D Itch Scale, Visual Analog Scale and KHemodialysis Comfort Scale -Version II.

Data collection forms will be applied twice in total, at the end of the 1st session (pretest) and at the end of the 8th session (posttest). The data obtained from the research will be analyzed in the Statistical Package for Social Science (SPSS) 21 statistical program. Variables covering the descriptive characteristics of the participants will be expressed in numbers and percentages. Whether the data has a normal distribution will be determined by the Kolmogrov Smirnov test and parametric and/or nonparametric tests will be used according to the results obtained. Statistical significance value will be accepted as p<.05.

DETAILED DESCRIPTION:
Hemodialysis treatment aims to increase the life expectancy and quality of life of individuals. However, it is known that hemodialysis, which is a life-preserving treatment, causes many undesirable problems in physical, psychological, social and economic areas, in addition to its targeted effects. Muscle cramps and itching are two of the most common symptoms during the hemodialysis treatment process, and it is known that all problems and symptoms encountered during the treatment process negatively affect the quality of life and comfort level of individuals. Management of symptoms experienced by individuals receiving hemodialysis treatment is very important due to their effects on both quality of life and comfort level. It is known that the effects of pharmacological treatments are limited in the management of symptoms encountered during the treatment process. Therefore, there is an increasing trend towards non-pharmacological methods in the management of these symptoms. Music therapy is one of the important complementary treatments preferred by nurses and is a method used to manage symptoms and has no side effects. With music therapy, physical, psychological, emotional and social well-being is increased by utilizing the therapeutic aspect of music.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Having been receiving hemodialysis treatment for at least 6 months,
* Being literate,
* Being open to collaboration,

Exclusion Criteria:

* Having sensory loss related to vision, hearing and communication,
* Having a psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Itch on the 5-D Itch Scale at Week 4 | Baseline and Week 4
  The 5-D Itch Scale is a reliable scale used to evaluate all causes of itching, including the duration, severity, course of itching, distribution in the body, and limitations caused by itching. On this scale, a total score of at least 5 points indicates no itching, and a maximum score of 25 points indicates very severe itching = (Week 4 Score- Baseline Score).
Change from Baseline in Muscle Cramps on the Visual Analog Scale at Week 4 | Baseline and Week 4
  Visual Analog Scale is a scale developed to convert some values that are difficult to measure numerically into numerical values. It is a scale evaluated on a horizontal line, divided into equal divisions of 10 cm, which includes the patient's impartial evaluation and indicates that one end is very good and the other end is very bad. The patient is asked to mark the number that best fits their symptoms. "0" represents the most comfortable situation, and "10" represents the worst situation = (Week 4 Score- Baseline Score).
Change from Baseline in Comfort on the Hemodialysis Comfort Scale -Version II at Week 4 | Baseline and Week 4
  Hemodialysis Comfort Scale -Version II consists of 26 items and is a five-point Likert type. The scale consists of six sub-dimensions: "physical relief, physical relaxation, psychospiritual relaxation, psychospiritual strengthening, environmental strengthening and sociocultural relief". The minimum score obtained from the scale is 26 and the highest score is 130. As the points received increase, the comfort of the patients also increases = (Week 4 Score- Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: soner telli, M.Sc., Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)